CLINICAL TRIAL: NCT06686277
Title: Effects Of Gong's Versus Mulligan Mobilization On Pain, Range Of Motion, Functional Disability and Quality Of Life In Patients With Adhesive Capsulitis
Brief Title: Effects Of Gong's Versus Mulligan Mobilization In Patients With Adhesive Capsulitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/24/0116
Record Dates: First submitted 2024-11-12; First posted 2024-11-13 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Adhesive Capsulitis of Shoulder
Keywords: Adhesive capsulitis; Functional Disability; Range of Motion
MeSH Terms: conditions — Bursitis

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial
Who Masked: Outcomes Assessor
Masking Description: Assessor blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gong's Technique Group (Experimental): The subject will sat on knee-high chair with the spine in a neutral position and comfortably extends both their arms. Therapist will stand on the side opposite to the affected side. The therapist will push the scapula of the affected side in a posterior to anterior direction with one hand, and pushed the humeral head in an anterior to posterior direction parallel to joint plane with the other hand. Simultaneously, the subject will quickly and powerfully perform shoulder abduction with elbow flexion and with palm facing inside and the back of the hand facing outside. During this time, the hands of the therapist kept facing the humeral head with long axis of the palm along with the long axis of the humerus. The therapist followed the subject performing shoulder abduction, at the same speed while maintaining a little distraction, and adding acceleration in the end range.
  Interventions: Other: Gong's Mobilization Technique
- Mulligan Mobilization (Experimental): For shoulder abduction, therapist applied a posterolateral gliding force over the head of the humerus, while patient actively abducted his arm. For shoulder flexion, the therapist applied a posterolateral glide as patient flexed his shoulder. For shoulder internal rotation, therapist applied an inferior shoulder glide and stabilized the scapula as the patient internally rotated his shoulder, and adducted his upper arm. As the therapist pushed the shoulder into adduction in this way, the head of the humerus was distracted laterally. Therapist hand in the axilla acted as a fulcrum.For shoulder external rotation,therapist applied posterolateral glide in sitting position
  Interventions: Other: Mulligan Mobilization Technique

INTERVENTIONS:
Other: Gong's Mobilization Technique — The therapist will push the scapula of the affected side in a posterior to anterior direction with one hand, and pushed the humeral head in an anterior to posterior direction parallel to joint plane with the other hand.
  Arms: Gong's Technique Group
Other: Mulligan Mobilization Technique — Mulligan Mobilization Technique
  Arms: Mulligan Mobilization

SUMMARY:
A Randomized Clinical Trial will be conducted at DHQ hospital kasur,BIT hospital kasur,Arif memorial hospital Lahore.Pre-diagnosed patients will be reassessed by applying (Shoulder Shrug Sign, Hand to neck, Hand to scapula, Hand to opposite scapula,Hand to back,Capsular pattern movement restriction)Plus all other special tests will be applied to confirm that symptoms are not due to other shoulder pathologies but are due to just adhesive capsulitis then through consecutive sampling technique on 60 patients they will be allocated using computer generated sampling(random number table) into Group A and Group B.

DETAILED DESCRIPTION:
A Randomized Clinical Trial will be conducted at DHQ hospital kasur,BIT hospital kasur,Arif memorial hospital Lahore.Pre-diagnosed patients will be reassessed by applying (Shoulder Shrug Sign, Hand to neck, Hand to scapula, Hand to opposite scapula,Hand to back,Capsular pattern movement restriction)Plus all other special tests will be applied to confirm that symptoms are not due to other shoulder pathologies but are due to just adhesive capsulitis then through consecutive sampling technique on 60 patients they will be allocated using computer generated sampling(random number table) into Group A and Group B. Group A will be treated with Gong's mobilization and Group B will be treated with Mulligan MWM The procedures will be performed Three sets of 10 repetitions, with 1 minute rest between sets,thrice per week for a total of six weeks. Pre and post intervention values will be taken on 1st day and after 6 weeks. Outcome measures will be conducted through VAS for pain,SPADI for functional disability , goniometer for range of motion ,SF-36 for quality of life after 6 weeks. Data will be analyzed during SPSS software version 25. After assessing normality of data by Shapiro-wilk test, it will be decided either parametric or non-parametric test will be used within a group or between two groups.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 to 50 years
* Both male and female
* Pre-diagnosed Unilateral Primary Frozen shoulder patients
* Prediagnosed Stage 3(Frozen phase) patients(27)

Exclusion Criteria:

* Patients with previous surgery in the shoulder joint
* History of recent fracture or severe trauma to the shoulder
* Diagnosed instability or previous history of dislocation
* Systemic inflammatory conditions(e.g.rheumatoid arthritis)

Ages: 40 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04-24 (Actual); Primary Completion 2025-01-24 (Estimated); Study Completion 2025-02-24 (Estimated)

PRIMARY OUTCOMES:
Level of Pain | Pre & Post 6 weeks
  Numeric Pain Rating Scale
Range of Motion | Pre & Post 6 weeks
  Goniometer
Functional Disability | Pre & Post 6 weeks
  Shoulder Pain and Disability Index
Quality of Life Level | Pre & Post 6 weeks
  Sort Form Survey-36

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Hassan, MSPT, Principal Investigator — Riphah International University
Locations (1):
- Iffat Anwar Medical Complex, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No